CLINICAL TRIAL: NCT06205433
Title: Evaluating the Impact of Training for IHSS Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Center for Caregiver Advancement (Unknown); Massachusetts Institute of Technology (Other); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2308001081
Record Dates: First submitted 2023-12-14; First posted 2024-01-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Home Care for Elderly or Disabled Individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHSS Basic Training (Experimental): Individuals in the treatment group will be invited to participate in CCA's IHSS Basic training program. The program is a 30 hour online course for IHSS providers, which teaches fundamental caregiving skills. Training includes personal care, infection control, nutrition and body mechanics, medication adherence, and home safety.
  Interventions: Other: IHSS Basic Training
- Control (No Intervention): No intervention is delivered to the control group. The control group will be unable to access CCA's training programs for two years following random assignment.

INTERVENTIONS:
Other: IHSS Basic Training — The intervention is the Center for Caregiver Advancements 30-hour IHSS Basic training course.
  Arms: IHSS Basic Training

SUMMARY:
This trial investigates whether high-quality training for consumer-directed home health workers impacts health outcomes for care consumers and employment outcomes for care workers. The investigators are conducting this study in the context of the In-Home Supportive Services (IHSS) program, a consumer-directed, Medicaid-funded home care program in California serving elderly and disabled Medicaid recipients. The investigators will partner with the Center for Caregiver Advancement (CCA), a training provider based in California, to conduct a randomized evaluation of the impact of training for IHSS workers on labor and health care outcomes. The evaluation will enroll IHSS workers in San Bernardino County, where CCA will be expanding its program.

Participants will be randomized to either a group that receives CCA's training or a control group that does not receive training.

Participants randomized to the training group will complete a 30 hour online course that teaches fundamental caregiving skills. Training includes personal care, infection control, nutrition and body mechanics, medication adherence, and home safety.

Researchers will compare outcomes between IHSS providers in the two groups and between IHSS consumers who receive care from the IHSS providers in the two groups to see if training impacts health, health care, and labor market outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current IHSS provider
* Live in San Bernardino County
* IHSS consumer lives in San Bernardino County

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of emergency department visits (for consumer) | 1 year after training begins

SECONDARY OUTCOMES:
Any emergency department visits (for consumer) | 1 year after training begins
Estimated annual health care spending (for consumer) | 1 year after training begins
  Estimated annual health care spending will be calculated by multiplying the number of inpatient admissions, emergency department visits, outpatient office visits, long term care stays, and prescription drugs by estimated average costs for those services among low income publicly insured adults.
Share of participants with falls resulting in a health care visit (for consumer) | 1 year after training begins
  The share of consumers with falls will be measured using diagnosis codes from medical claims
Share of participants with urinary tract infections resulting in a health care visit (for consumer) | 1 year after training begins
  The share of consumers with urinary tract infections will be measured using diagnosis codes from medical claims
Share of participants with pressure ulcers resulting in a health care visit (for consumer) | 1 year after training begins
  The share of consumers with pressure ulcers will be measured using diagnosis codes from medical claims
Share of participants with nursing facility utilization (for consumer) | 1 year after training begins
  The share of consumers who have a stay in a skilled nursing facility, rehab, or long term care facility during the year after training begins.
Share of participants still employed in IHSS (for provider) | 1 year after training begins
  The share of IHSS provider participants who remain as workers in the IHSS program 1 year after the start of training.
Caregiving knowledge (for provider) | 0-3 months after completion of training
  Proportion of correct answers out of 18 true false knowledge questions
Total length of stay in nursing facilities (for consumer) | 1 year after training begins
  The number of days spent per consumer in a skilled nursing facility, rehab, or long term care facility during the year after training begins.
IHSS earnings (for provider) | 1 year after training begins
  IHSS earnings for providers, measured weekly, quarterly, and annually, drawn from IHSS payroll data
IHSS hours worked (for provider) | 1 year after training begins
  IHSS hours worked for providers, measured weekly, quarterly, and annually, drawn from IHSS payroll data

OTHER OUTCOMES:
Any hospital admissions (for consumer) | 1 year after training begins
Number of hospital admissions (for consumer) | 1 year after training begins
Total length of stay in hospital (for consumer) | 1 year after training begins
Depression (for provider) | 0-3 months after completion of training
  Patient Health Questionnaire-2 (PHQ-2). Scores range from 0 to 6, with higher values indicating worse outcomes. A score of 3 or higher identifies possible cases of major depressive disorder.
Anxiety (for provider) | 0-3 months after completion of training
  Generalized Anxiety Disorder 2-item (GAD-2). Scores range from 0 to 6, with higher values indicating worse outcomes. A score of 3 or higher identifies possible cases of generalized anxiety disorder.
Caregiver wellbeing (for provider) | 0-3 months after completion of training
  18 question caregiver self assessment questionnaire developed by the American Medical Association (https://www.healthinaging.org/tools-and-tips/caregiver-self-assessment-questionnaire). Includes 16 Yes/No questions and 2 scale of 1 to 10 questions, with higher values indicating worse outcomes. 10 or more yes answers, having crying spells, feeling completely overwhelmed, a stress rating of >=6 out of 10, or health rating of >= 6 out of 10 all indicate distress.
Caregiver job satisfaction (for provider) | 0-3 months after completion of training
  Self-reported answer to "Overall, how satisfied are you with your IHSS job?" on a 5-point Likert scale from very dissatisfied to very satisfied
Number of consumers served (for provider) | 1 year after training begins
  How many people the provider is paid to care for as part of the IHSS program

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Notowidigdo, PhD, Principal Investigator — University of Chicago; David Autor, Phd, Principal Investigator — Massachusetts Institute of Technology; Amy Finkelstein, PhD, Principal Investigator — Massachusetts Institute of Technology; Anna Russo, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- San Bernardino County, San Bernardino, California, United States

IPD SHARING:
Plan to Share IPD: Yes
To the extent allowed by our data use agreements with administrative data providers, we will share de-identified data and analysis code at the conclusion of the project.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available after publication and will be hosted on a public research data repository such as the Harvard Dataverse (dataverse.org).